CLINICAL TRIAL: NCT02478632
Title: An Evaluation of Bone Mineral Density in HIV-1-infected Adult Subjects Switching From a Tenofovir-containing Antiretroviral Therapy Regimen to a Dolutegravir Plus Rilpivirine Regimen
Brief Title: Bone Mineral Density in Human Immunodeficiency Virus Type 1 (HIV-1)-Infected Adult Subjects Switching From a Tenofovir Regimen to a Dolutegravir Plus Rilpivirine Regimen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Janssen Pharmaceuticals (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202094
Record Dates: First submitted 2015-05-28; First posted 2015-06-23 (Estimated); Results first posted 2017-10-20 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: HIV Infections
Keywords: tenofovir disoproxil fumarate; dolutegravir plus rilpivirine; two-drug regimen; bone mineral density; dual energy X-ray absorptiometry (DEXA); Human Immunodeficiency Virus-1; nucleoside reverse transcriptase inhibitor -sparing regimen; integrase inhibitor
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CAR (Active Comparator): Participants do not receive study medication in this study 202094. Participants group carried over from the parent study 201636 (SWORD-1) or 201637 (SWORD-2).
  Interventions: Drug: Subjects do not receive study medication in this study 202094
- DTG 50 mg + RPV 25 mg (Experimental): Participants do not receive study medication in this study 202094. Participants group carried over from the parent study 201636 (SWORD-1) or 201637 (SWORD-2)
  Interventions: Drug: Subjects do not receive study medication in this study 202094

INTERVENTIONS:
Drug: Subjects do not receive study medication in this study 202094 — Participants do not receive study medication in this study 202094.

SUMMARY:
The purpose of this study is to evaluate any change from baseline in bone mineral density (BMD) in subjects following the switch from a triple antiretroviral therapy (ART) regimen containing Tenofovir disoproxil fumarate (TDF) to the nucleoside reverse transcriptase inhibitor (NRTI) - sparing two - drug regimen of dolutegravir (DTG) + rilpivirine (RPV) in subjects participating in the parent studies 201636 and 201637 (SWORD-1 and SWORD-2).

This open-label, parallel group, study is a sub-study which will recruit subjects who are receiving ART regimens which include TDF at the time of randomization to receive treatment in one of two identical parent studies 201636 and 201637 (SWORD-1 and SWORD-2). These are Phase III, randomised, open-label, multicentre, parallel-group, non-inferiority studies evaluating the efficacy, safety, and tolerability of switching to DTG plus RPV from current integrase inhibitor (INI)-, non NNRTI-, or protease inhibitor (PI)-based antiretroviral regimen in HIV-1-infected adults who are virologically suppressed, having HIV-1 ribonucleic acid (RNA) levels <50 copies per millilitre (c/mL). Randomisation in the parent studies will be stratified by baseline third agent class (INI, NNRTI, or PI), age group (< or =>50 years old) and participation in this Dual energy X-ray absorptiometry (DEXA) sub-study, therefore there will also be balance across the treatment arms in this sub-study both overall and with respect to baseline third agent class and age at entry.

The study population will include approximately 75 evaluable subjects recruited from the Early Switch DTG + RPV treatment group of the parent studies 201636 and 201637, and approximately 75 evaluable subjects from the Late Switch group who continue their current antiretroviral therapy (CAR) through to Week 52 across both the 201636 and 201637 (SWORD-1 and SWORD-2) studies. Subjects participating in study 202094 will have DEXA scans performed at Day 1 and at study Weeks 48, 100 and 148 in parallel with the corresponding scheduled visits in the parent studies.

ELIGIBILITY:
Inclusion Criteria:

* Screened and eligible but not yet randomised to either of the parent studies 201636 (SWORD-1) or 201637 (SWORD-2)
* Receiving an ART regimen which contains TDF
* Female subjects of child bearing potential with a negative pregnancy test at both Screening and Day 1 and agrees to use one of the methods of contraception described in the protocols of the parent studies 201636 (SWORD-1) and 201637 (SWORD-2) to avoid pregnancy. Any contraception method must be used consistently, throughout the study period in accordance with the approved product label, including adherence to appropriate 'run in' periods for hormonal contraception
* Subject is willing and able to understand the requirements of study participation and provide signed and dated written informed consent prior to Screening. Subject is considered an appropriate candidate for participation in this study
* For subjects enrolled in France: a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category

Exclusion Criteria:

* Less than three vertebra in the range of L1 to L4 that are suitable for BMD measurement by DEXA scan
* Bilateral hip replacement
* Uncontrolled thyroid disease: thyroid stimulating hormone (TSH) above normal range, and considered to indicate a requirement for thyroid replacement therapy
* Male hypogonadism: serum testosterone < 300 nanogram per decilitre (ng/dL) on a sample collected before 10:00 in the morning and the subject is able and willing to start testosterone replacement therapy
* Endocrine diseases including Cushing's syndrome and diabetes mellitus
* History of fragility fractures
* Ever treated for osteoporosis with bisphosphonates, oestrogen receptor modulators or other therapies, and / or severe osteoporosis as indicated by a prior DEXA scan derived T-score of -3.5 or lower value
* Body mass index (BMI) < 18 kilogram per meter (kg/m)^2 or =>40 kg/m^2
* Vitamin D deficiency: 25 Hydroxy Vitamin D < 15ng/mL
* Any pre-existing physical or mental condition (including substance abuse disorder) which, in the opinion of the investigator, may interfere with the subject's ability to comply with the scheduled protocol evaluations or which may compromise the safety of the subject
* Current use or intent to initiate, tamoxifen, bone-related treatment, e.g. biphosphonates, osteoporosis medications including selective oestrogen receptor modulator medicines (raloxifene, arzoxifene and lasofoxifene), growth hormone or anabolic steroids, except for testosterone as specified below, during the study period
* The following are excluded unless they have been given for at least 6 months prior to Day 1, and there is no plan to stop them during the study: Anti-convulsant therapy and hormonal therapy, including female hormone replacement therapy or testosterone as a replacement therapy or supplement
* Women who are pregnant, breastfeeding or who plan to become pregnant or breast feed during the study period
* Subject enrolled, or anticipated to be selected to participate following study registration, in an investigational clinical protocol/s in addition to one of the parent studies 201636 or 201637 (SWORD-1 or SWORD-2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-06-12 (Actual); Primary Completion 2016-09-16 (Actual); Study Completion 2018-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (28):
- United States (7):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Lynchburg, Virginia
- Argentina (4):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Ciudad de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
- Belgium (3):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Liège
- Canada (4):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec
- Spain (9):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Cartagena (Murcia)
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Seville
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20273

REFERENCES:
- [Background] McComsey GA, Lupo S, Parks D, Poggio MC, De Wet J, Kahl LP, Angelis K, Wynne B, Vandermeulen K, Gartland M, Cupo M, Aboud M; 202094 Sub-Study Investigators. Switch from tenofovir disoproxil fumarate combination to dolutegravir with rilpivirine improves parameters of bone health. AIDS. 2018 Feb 20;32(4):477-485. doi: 10.1097/QAD.0000000000001725. PMID 29239893

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants from early switch dolutegravir (DTG) plus rilpivirine (RPV) treatment groups and from late switch group who continue their current antiretroviral regimen (CAR) through Week 52 across both NCT02429791 and NCT02422797 were included in this sub-study 202094.
Pre-assignment Details: Total 146 participants were screened, of which, 44 were screen failures and 102 were registered to study 202094. The study included an early switch phase and a late switch phase.
Groups:
- DTG + RPV: Participants received randomized DTG together with RPV once daily in an open-label fashion up to Week 52 during early switch phase in the parent study and continued to receive DTG + RPV up to Week 148 during the late switch phase in the parent study (study medication was administered in the parent study and not in study 202094).
- Current Antiretroviral Regimen: Participants continued to receive their current antiretroviral regimen (CAR) (two nucleoside reverse transcriptase inhibitors [NRTIs] + a third agent). A third agent included either an: integrase strand transfer inhibitor (INSTI), a non-nucleoside reverse transcriptase inhibitor (NNRTI) or a protease inhibitor (PI). CAR was administered according to the approved labeling in an open-label fashion up to Week 52 during early switch phase in the parent study. At Week 52, participants with human immunodeficiency virus-1 (HIV-1) ribonucleic acid (RNA) <50 copies per milliliter (c/mL), switched to DTG + RPV once daily and were followed until Week 148 in the parent study (study medication was administered in the parent study and not in study 202094).
Period: Early Switch Phase (Up to Week 52)
Arm/Group | DTG + RPV | Current Antiretroviral Regimen
Started | 53 | 49
Completed | 49 | 44
Not Completed | 4 | 5
Not completed — Withdrawal from parent study | 4 | 5
Period: Late Switch Phase (Week 52 to Week 148)
Arm/Group | DTG + RPV | Current Antiretroviral Regimen
Started | 49 | 44
Completed | 42 | 40
Not Completed | 7 | 4
Not completed — Withdrawal from parent study | 2 | 3
Not completed — Prohibited medication use | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DTG + RPV | Current Antiretroviral Regimen | Total
Number analyzed (Participants) | 53 | 49 | 102
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.6 (10.80) | 44.8 (10.66) | 43.7 (10.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 26 | 53
  Male | 26 | 23 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/ Alaska native Heritage | 4 | 1 | 5
  Asian- Central/South Asian Heritage | 0 | 1 | 1
  Asian- Japanese/East Asian (EA)/ South EA heritage | 2 | 0 | 2
  Black / African American | 3 | 7 | 10
  White | 44 | 40 | 84

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Total Hip Bone Mineral Density (BMD) at Week 48
Description: Percent change in BMD (expressed as areal density in grams per centimeter square [g/cm^2]) as specified by dual energy X-ray absorptiometry (DEXA) scans of the left 'total hip' which included the femoral neck, trochanter and inter-trochanter areas was assessed by areal density at Baseline and Week 48. The estimated value in the statistical analysis is this difference and the upper and lower limit values shown are the 95% confidence intervals. Baseline was considered as Day 1 and percent change from Baseline was calculated as Value at Week 48 minus Baseline value divided by Baseline value multiplied by 100. An analysis of covariance (ANCOVA) model was used to compare the difference. The analysis was performed on Intent-to-Treat exposed DEXA (ITT-ED) Population which comprised of all participants in the ITT-E Population who received at least one dose of study treatment, and who were registered for the 202094 study.
Time Frame: Baseline (Day 1) and Week 48
Population: ITT-ED Population. Only those participants with data available at specified time point were analyzed.
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | DTG + RPV | Current Antiretroviral Regimen
Number analyzed (Participants) | 46 | 35
Percent change | 1.34 [0.68 to 2.01] | 0.05 [-0.71 to 0.82]
Statistical Analysis 1: Comparison: DTG + RPV vs Current Antiretroviral Regimen; Test type: Superiority; p = 0.014, ANCOVA; Mean Difference (Final Values) = 1.29, 95% CI 2-sided [0.27 to 2.31]

2. Secondary Outcome: Percent Change From Baseline in Lumbar Spine BMD at Week 48
Description: Percent change in BMD (expressed as areal density in g/cm^2) as specified by DEXA scans of the 'lumbar spine' which included the first lumbar vertebra (L1) to the fourth lumbar vertebra (L4) was assessed by areal density at Baseline and Week 48. The difference is adjusted percent change from Baseline to Week 48 between treatment groups. The estimated value in the statistical analysis is this difference and the upper and lower limit values shown are the 95% confidence intervals. Baseline was considered as Day 1 value and percent change from Baseline was calculated as Value at Week 48 minus Baseline value divided by Baseline value multiplied by 100. An ANCOVA model was used to compare the difference in percentage change from Baseline at week 48 in lumbar spine BMD between the DTG+RPV and CAR arms.
Time Frame: Baseline (Day 1) and Week 48
Population: ITT-ED Population. Only those participants with data available at specified time point were analyzed.
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | DTG + RPV | Current Antiretroviral Regimen
Number analyzed (Participants) | 46 | 35
Percent change | 1.46 [0.65 to 2.28] | 0.15 [-0.79 to 1.09]
Statistical Analysis 1: Comparison: DTG + RPV vs Current Antiretroviral Regimen; Test type: Superiority; p = 0.039, ANCOVA; Mean Difference (Final Values) = 1.32, 95% CI 2-sided [0.07 to 2.57]

3. Secondary Outcome: Percent Change From Baseline in Total Hip and Lumbar Spine BMD-DTG+RPV Early Switch Group Through Early and Late Switch Phase
Description: Percent change in BMD (expressed as areal density in g/cm^2) as specified by DEXA scans of left 'total hip' which included femoral neck, trochanter and inter-trochanter areas and 'lumbar spine' which included L1 to L4 was assessed by areal density. Percent change from Baseline is post-dose value minus Baseline value divided by Baseline value multiplied by 100. BMD parameters at Weeks 48, 100 and 148 reflect data adjusted following the ongoing longitudinal and cross-calibration of multiple DEXA scanner instruments in this study. Data presented through Week 48 only represent results of Week 48 Primary Endpoint analysis which applied DEXA scanner calibrations though Week 48, with no subsequent calibration applied. In the final analysis conducted at Week 148, DEXA scanner calibration data acquired from Day 1 to Week 148 was applied to all raw DEXA BMD data at Weeks 48, 100 and 148. Hence, actual values of Week 48 DEXA data may vary slightly between Weeks 48 and 148 analyses.
Time Frame: Baseline (Day 1), Week 48, Week 100 and Week 148
Population: ITT-ED Population. Only those participants with data available at specified time point were analyzed (represented by n=X) in category titles.
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | DTG + RPV
Number analyzed (Participants) | 53
Percent change
  Total hip; Week 48; n=46: number analyzed (Participants) | 46
  Total hip; Week 48; n=46 | 1.492 [0.74 to 2.24]
  Total hip; Week 100; n=41: number analyzed (Participants) | 41
  Total hip; Week 100; n=41 | 1.081 [0.06 to 2.10]
  Total hip; Week 148; n=40: number analyzed (Participants) | 40
  Total hip; Week 148; n=40 | 0.978 [-0.23 to 2.18]
  Lumbar spine; Week 48; n=46: number analyzed (Participants) | 46
  Lumbar spine; Week 48; n=46 | 1.648 [0.83 to 2.46]
  Lumbar spine; Week 100; n=43: number analyzed (Participants) | 43
  Lumbar spine; Week 100; n=43 | 0.810 [-0.39 to 2.01]
  Lumbar spine; Week 148; n=42: number analyzed (Participants) | 42
  Lumbar spine; Week 148; n=42 | 0.526 [-0.93 to 1.98]

4. Secondary Outcome: Percent Change From Late Switch (LS) Baseline (Week 48) Through Week 148 in Total Hip and Lumbar Spine BMD-CAR Late Switch Group Through Late Switch Phase
Description: Percent change in BMD (expressed as areal density in g/cm^2) as specified by DEXA scans of the left 'total hip' which included the femoral neck, trochanter and inter-trochanter areas was assessed by areal density at indicated time points. Percent change in BMD as specified by DEXA scans of the 'lumbar spine' which included the first lumbar vertebra (L1) to the fourth lumbar vertebra (L4) was assessed by areal density at indicated time points. The last pre-switch value (Week 48) was considered as LS Baseline and percent change from LS Baseline was calculated as post-dose visit value minus LS Baseline value divided by LS Baseline value multiplied by 100. The analysis was based on Late-Switch Intent-to-Treat Exposed DEXA (LS-ITT-ED) Population which comprised of all participants in the LS-ITT-E Population, and who were registered for the DEXA study.
Time Frame: LS Baseline (Week 48), Week 100 and Week 148
Population: LS ITT-ED Population. Only those participants with data available at specified time point were analyzed (represented by n=X) in category titles.
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Current Antiretroviral Regimen
Number analyzed (Participants) | 44
Percent change
  Total hip; Week 100; n=41: number analyzed (Participants) | 41
  Total hip; Week 100; n=41 | 1.107 [0.25 to 1.96]
  Total hip; Week 148; n=40: number analyzed (Participants) | 40
  Total hip; Week 148; n=40 | 1.275 [0.39 to 2.16]
  Lumbar spine; Week 100; n=41: number analyzed (Participants) | 41
  Lumbar spine; Week 100; n=41 | 1.135 [0.11 to 2.16]
  Lumbar spine; Week 148; n=40: number analyzed (Participants) | 40
  Lumbar spine; Week 148; n=40 | 0.436 [-0.64 to 1.51]

5. Secondary Outcome: Change From Baseline in Total Hip and Lumbar Spine BMD at Week 48 Assessed by T-score and Z-score
Description: Total hip and lumbar spine BMD was assessed by T-scores and Z-scores. Day 1 was considered as Baseline. Change from Baseline was calculated as the value at Week 48 minus Baseline. DEXA scans of the left 'total hip' (femoral neck, hip, inter-trochanter areas, trochanter) and 'lumbar spine' (lumbar vertebral column) were performed. T-score is the number of standard deviations above or below the mean BMD of a 30-year-old participant of the same sex. Caucasian reference values were used for all participants to calculate T-scores. T-score values > -1.0 are considered normal, T-score values <= -1.0 to > -2.5 indicate osteopenia, T-score values <= -2.5 to <-3.5 indicate osteoporosis and T-score values <= -3.5 indicate severe osteoporosis. The Z-score is the number of standard deviations above or below the mean BMD for a reference population of same age and sex and in this study. Caucasian reference values were used in calculation of Z-scores.
Time Frame: Baseline (Day 1) and Week 48
Population: ITT-ED Population. Only those participants with data available at specified time point were analyzed.
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | DTG + RPV | Current Antiretroviral Regimen
Number analyzed (Participants) | 46 | 35
Scores on a scale
  Total hip; T-score | 0.09 [0.05 to 0.14] | 0.01 [-0.05 to 0.06]
  Total hip; Z-score | 0.11 [0.06 to 0.15] | 0.02 [-0.03 to 0.08]
  Lumbar spine; T-score | 0.13 [0.05 to 0.20] | 0.01 [-0.08 to 0.10]
  Lumbar spine; Z-score | 0.17 [0.09 to 0.25] | 0.02 [-0.07 to 0.11]
Statistical Analysis 1: Comparison: DTG + RPV vs Current Antiretroviral Regimen; Test type: Superiority; p = 0.016, ANCOVA — p value for the difference in adjusted change from Baseline at Week 48 in total hip T-scores between the DTG+RPV and CAR groups; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [0.02 to 0.16] — The analysis estimated the difference between DTG+RPV and CAR in total hip T-scores
Statistical Analysis 2: Comparison: DTG + RPV vs Current Antiretroviral Regimen; Test type: Superiority; p = 0.026, ANCOVA — p value for the difference in adjusted change from Baseline at Week 48 in total hip Z-scores between the DTG+RPV and CAR groups; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [0.01 to 0.15] — The analysis estimated difference between DTG+RPV and CAR in total hip Z-score
Statistical Analysis 3: Comparison: DTG + RPV vs Current Antiretroviral Regimen; Test type: Superiority; p = 0.049, ANCOVA — p value for the difference in adjusted change from Baseline at Week 48 in lumbar spine T-scores between the DTG+RPV and CAR groups; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [0.00 to 0.23] — The analysis estimated difference between DTG+RPV and CAR for lumbar spine T-score
Statistical Analysis 4: Comparison: DTG + RPV vs Current Antiretroviral Regimen; Test type: Superiority; p = 0.013, ANCOVA — p value for the difference in adjusted change from Baseline at Week 48 in lumbar spine Z-scores between the DTG+RPV and CAR groups; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [0.03 to 0.27] — The analysis estimated difference between DTG+RPV and CAR in lumbar spine Z-score

6. Secondary Outcome: Change From Baseline in Total Hip and Lumbar Spine BMD as Assessed by T-scores and Z-scores - DTG+RPV Early Switch Group Through Early and Late Switch Phase
Description: T-score is the number of standard deviations above or below the mean BMD of a 30-year-old participant of same sex. Caucasian reference values were used to calculate T- and Z- scores. T-score values: > -1.0 is normal; <= -1.0 to > -2.5 indicate osteopenia; <= -2.5 to <-3.5 indicate osteoporosis; <= -3.5 indicate severe osteoporosis. Z-score is the number of standard deviations above or below the mean BMD for a reference population of same age and sex in this study. Change from Baseline is post-dose visit value minus Baseline value. Data for Week 48 only represent final results of Week 48 Primary Endpoint analysis which applied DEXA scanner calibrations through Week 48, with no subsequent calibration applied. In the final analysis conducted at Week 148, DEXA scanner calibration data acquired from Day 1 to Week 148 was applied to all raw DEXA BMD data at Weeks 48, 100 and 148. Hence, actual values of Week 48 DEXA data may vary slightly between Weeks 48 and 148 analyses.
Time Frame: Baseline (Day 1), Week 48, Week 100 and Week 148
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | DTG + RPV
Number analyzed (Participants) | 53
Scores on a scale
  Total hip; T-score; Week 48; n=46: number analyzed (Participants) | 46
  Total hip; T-score; Week 48; n=46 | 0.101 (0.1681)
  Total hip; T-score; Week 100; n=41: number analyzed (Participants) | 41
  Total hip; T-score; Week 100; n=41 | 0.066 (0.2248)
  Total hip; T-score; Week 148; n=40: number analyzed (Participants) | 40
  Total hip; T-score; Week 148; n=40 | 0.062 (0.2600)
  Total hip; Z-score; Week 48; n=46: number analyzed (Participants) | 46
  Total hip; Z-score; Week 48; n=46 | 0.115 (0.1742)
  Total hip; Z-score; Week 100; n=41: number analyzed (Participants) | 41
  Total hip; Z-score; Week 100; n=41 | 0.107 (0.2222)
  Total hip; Z-score; Week 148; n=40: number analyzed (Participants) | 40
  Total hip; Z-score; Week 148; n=40 | 0.117 (0.2757)
  Lumbar spine; T-score; Week 48; n=46: number analyzed (Participants) | 46
  Lumbar spine; T-score; Week 48; n=46 | 0.139 (0.2511)
  Lumbar spine; T-score; Week 100; n=43: number analyzed (Participants) | 43
  Lumbar spine; T-score; Week 100; n=43 | 0.059 (0.3510)
  Lumbar spine; T-score; Week 148; n=42: number analyzed (Participants) | 42
  Lumbar spine; T-score; Week 148; n=42 | 0.034 (0.4183)
  Lumbar spine; Z-score; Week 48; n=46: number analyzed (Participants) | 46
  Lumbar spine; Z-score; Week 48; n=46 | 0.182 (0.2563)
  Lumbar spine; Z-score; Week 100; n=43: number analyzed (Participants) | 43
  Lumbar spine; Z-score; Week 100; n=43 | 0.142 (0.3868)
  Lumbar spine; Z-score; Week 148; n=42: number analyzed (Participants) | 42
  Lumbar spine; Z-score; Week 148; n=42 | 0.139 (0.4507)

7. Secondary Outcome: Change From LS Baseline (Week 48) Through Week 148 in Total Hip and Lumbar Spine BMD as Assessed by T-scores and Z-scores-CAR Late Switch Group Through Late Switch Phase
Description: The last pre-switch value (Week 48) was considered as LS Baseline and change from LS Baseline was calculated as the post-dose visit value minus LS Baseline value. DEXA scans of the left 'total hip' (femoral neck, hip, inter-trochanter areas, trochanter) and 'lumbar spine' (lumbar vertebral column) were performed. T-score is the number of standard deviations above or below the mean BMD of a 30-year-old participant of the same sex. Caucasian reference values were used for all participants to calculate T-scores. T-score values > -1.0 are considered normal, T-score values <= -1.0 to > -2.5 indicate osteopenia, T-score values <= -2.5 to <-3.5 indicate osteoporosis and T-score values <= -3.5 indicate severe osteoporosis. The Z-score is the number of standard deviations above or below the mean BMD for a reference population of same age and sex and in this study. Caucasian reference values were used in calculation of Z-scores.
Time Frame: LS Baseline (Week 48), Week 100, Week 148
Population: LS ITT-ED Population. Only those participants with data available at specified time point were analyzed (represented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Current Antiretroviral Regimen
Number analyzed (Participants) | 44
Scores on a scale
  Total hip; T-score; Week 100; n=41: number analyzed (Participants) | 41
  Total hip; T-score; Week 100; n=41 | 0.080 (0.1957)
  Total hip; T-score; Week 148; n=40: number analyzed (Participants) | 40
  Total hip; T-score; Week 148; n=40 | 0.091 (0.1995)
  Total hip; Z-score; Week 100; n=41: number analyzed (Participants) | 41
  Total hip; Z-score; Week 100; n=41 | 0.107 (0.2055)
  Total hip; Z-score; Week 148; n=40: number analyzed (Participants) | 40
  Total hip; Z-score; Week 148; n=40 | 0.125 (0.2117)
  Lumbar spine; T-score; Week 100; n=41: number analyzed (Participants) | 41
  Lumbar spine; T-score; Week 100; n=41 | 0.111 (0.2914)
  Lumbar spine; T-score; Week 148; n=40: number analyzed (Participants) | 40
  Lumbar spine; T-score; Week 148; n=40 | 0.049 (0.3204)
  Lumbar spine; Z-score; Week 100; n=41: number analyzed (Participants) | 41
  Lumbar spine; Z-score; Week 100; n=41 | 0.176 (0.2598)
  Lumbar spine; Z-score; Week 148; n=40: number analyzed (Participants) | 40
  Lumbar spine; Z-score; Week 148; n=40 | 0.127 (0.3392)

8. Secondary Outcome: Percent Change From Baseline in Total Hip and Lumbar Spine BMD at Week 48 by Baseline Third Agent
Description: Total hip and lumbar spine BMD (expressed as areal density in g/cm^2) assessed by third agent class (INSTI, NNRTI, PI) at indicated time points. Percent change from Baseline was calculated as value at Week 48 minus Baseline value divided by Baseline value multiplied by 100. Value at Day 1 was considered as Baseline. An ANCOVA model adjusted for Baseline BMD values was used to compare the difference in percent change from Baseline to Week 48 in total hip BMD or in lumbar spine BMD between the DTG+RPV and CAR arms by third agent class: INSTI, NNRTI or PI.
Time Frame: Baseline (Day 1) and Week 48
Population: ITT-ED Population. Only those participants with data available at specified time point were analyzed (represented by n=X in category titles).
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | DTG + RPV | Current Antiretroviral Regimen
Number analyzed (Participants) | 46 | 35
Percent change
  Total hip; INSTI; n=7, 4: number analyzed (Participants) | 7 | 4
  Total hip; INSTI; n=7, 4 | 2.03 [-0.47 to 4.53] | 1.38 [-1.93 to 4.69]
  Total hip; NNRTI; n=28, 24: number analyzed (Participants) | 28 | 24
  Total hip; NNRTI; n=28, 24 | 1.33 [0.51 to 2.16] | -0.27 [-1.16 to 0.62]
  Total hip; PI; n=11, 7: number analyzed (Participants) | 11 | 7
  Total hip; PI; n=11, 7 | 1.11 [-0.34 to 2.56] | 0.12 [-1.72 to 1.95]
  Lumbar spine; INSTI; n=7, 3: number analyzed (Participants) | 7 | 3
  Lumbar spine; INSTI; n=7, 3 | 1.43 [-0.31 to 3.17] | -2.42 [-5.08 to 0.24]
  Lumbar spine; NNRTI; n=28, 26: number analyzed (Participants) | 28 | 26
  Lumbar spine; NNRTI; n=28, 26 | 1.38 [0.34 to 2.42] | 0.12 [-0.96 to 1.20]
  Lumbar spine; PI; n=11, 6: number analyzed (Participants) | 11 | 6
  Lumbar spine; PI; n=11, 6 | 1.78 [-0.22 to 3.78] | 1.40 [-1.32 to 4.11]
Statistical Analysis 1: Comparison: DTG + RPV vs Current Antiretroviral Regimen; Test type: Other; Mean Difference (Final Values) = 0.65, 95% CI 2-sided [-3.51 to 4.81] — The analysis refers to INSTI and total hip
Statistical Analysis 2: Comparison: DTG + RPV vs Current Antiretroviral Regimen; Test type: Other; Mean Difference (Final Values) = 1.60, 95% CI 2-sided [0.39 to 2.81] — The analysis refers to NNRTI and total hip
Statistical Analysis 3: Comparison: DTG + RPV vs Current Antiretroviral Regimen; Test type: Other; Mean Difference (Final Values) = 1.00, 95% CI 2-sided [-1.39 to 3.38] — this analysis refers to PI and total hip
Statistical Analysis 4: Comparison: DTG + RPV vs Current Antiretroviral Regimen; Test type: Other; Mean Difference (Final Values) = 3.85, 95% CI 2-sided [0.67 to 7.03] — this analysis refers to INSTI and lumbar spine
Statistical Analysis 5: Comparison: DTG + RPV vs Current Antiretroviral Regimen; Test type: Other; Mean Difference (Final Values) = 1.25, 95% CI 2-sided [-0.26 to 2.76] — this analysis refers to NNRTI and lumbar spine
Statistical Analysis 6: Comparison: DTG + RPV vs Current Antiretroviral Regimen; Test type: Other; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [-3.00 to 3.77] — this analysis refers to PI and lumbar spine

9. Secondary Outcome: Change From Baseline in Total Hip and Lumbar Spine BMD T-scores and Z-scores at Week 48 by Baseline Third Agent
Description: Total hip and lumbar spine BMD was assessed by Baseline third agent class (INSTI, NNRTI, PI) using T-scores and Z-scores at Baseline and Week 48. DEXA scans of hip and spine were performed. Value at Day 1 was considered as Baseline. Change from Baseline was calculated as the value at Week 48 minus Baseline value. T-score is the number of standard deviations above or below the mean BMD of a 30-year-old participant of the same sex. Caucasian reference values were used for all participants to calculate T-scores. T-score values > -1.0 are considered normal, T-score values <= -1.0 to > -2.5 indicate osteopenia, T-score values <= -2.5 to <-3.5 indicate osteoporosis and T-score values <= -3.5 indicate severe osteoporosis. The Z-score is the number of standard deviations above or below the mean BMD for a reference population of same age and sex and in this study. Caucasian reference values were used in calculation of Z-scores.
Time Frame: Baseline (Day 1) and Week 48
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | DTG + RPV | Current Antiretroviral Regimen
Number analyzed (Participants) | 46 | 35
Scores on a scale
  Total hip; T-score; INSTI; n=7, 4: number analyzed (Participants) | 7 | 4
  Total hip; T-score; INSTI; n=7, 4 | 0.13 [-0.04 to 0.29] | 0.11 [-0.11 to 0.33]
  Total hip; T-score; NNRTI; n=28, 24: number analyzed (Participants) | 28 | 24
  Total hip; T-score; NNRTI; n=28, 24 | 0.09 [0.04 to 0.15] | -0.02 [-0.08 to 0.04]
  Total hip; T-score; PI; n=11, 7: number analyzed (Participants) | 11 | 7
  Total hip; T-score; PI; n=11, 7 | 0.08 [-0.02 to 0.18] | 0.01 [-0.12 to 0.13]
  Total hip; Z-score; INSTI; n=7, 4: number analyzed (Participants) | 7 | 4
  Total hip; Z-score; INSTI; n=7, 4 | 0.18 [-0.00 to 0.36] | 0.12 [-0.13 to 0.36]
  Total hip; Z-score; NNRTI; n=28, 24: number analyzed (Participants) | 28 | 24
  Total hip; Z-score; NNRTI; n=28, 24 | 0.10 [0.04 to 0.16] | 0.00 [-0.06 to 0.06]
  Total hip; Z-score; PI; n=11, 7: number analyzed (Participants) | 11 | 7
  Total hip; Z-score; PI; n=11, 7 | 0.08 [-0.02 to 0.19] | 0.05 [-0.08 to 0.18]
  Lumbar spine; T-score; INSTI; n=7, 3: number analyzed (Participants) | 7 | 3
  Lumbar spine; T-score; INSTI; n=7, 3 | 0.14 [-0.04 to 0.33] | -0.22 [-0.51 to 0.07]
  Lumbar spine; T-score; NNRTI; n=28, 26: number analyzed (Participants) | 28 | 26
  Lumbar spine; T-score; NNRTI; n=28, 26 | 0.11 [0.02 to 0.21] | 0.00 [-0.10 to 0.10]
  Lumbar spine; T-score; PI; n=11, 6: number analyzed (Participants) | 11 | 6
  Lumbar spine; T-score; PI; n=11, 6 | 0.15 [-0.03 to 0.34] | 0.14 [-0.11 to 0.39]
  Lumbar spine; Z-score; INSTI; n=7, 3: number analyzed (Participants) | 7 | 3
  Lumbar spine; Z-score; INSTI; n=7, 3 | 0.19 [0.01 to 0.38] | -0.19 [-0.48 to 0.10]
  Lumbar spine; Z-score; NNRTI; n=28, 26: number analyzed (Participants) | 28 | 26
  Lumbar spine; Z-score; NNRTI; n=28, 26 | 0.13 [0.04 to 0.23] | 0.01 [-0.09 to 0.11]
  Lumbar spine; Z-score; PI; n=11,6: number analyzed (Participants) | 11 | 6
  Lumbar spine; Z-score; PI; n=11,6 | 0.24 [0.06 to 0.41] | 0.19 [-0.05 to 0.43]
Statistical Analysis 1: Comparison: DTG + RPV vs Current Antiretroviral Regimen; Test type: Other; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.26 to 0.30] — The analysis estimated comparison of change from baseline to Week 48 between the DTG+RPV and CAR groups in total hip T-scores by baseline third agent INSTI
Statistical Analysis 2: Comparison: DTG + RPV vs Current Antiretroviral Regimen; Test type: Other; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [0.03 to 0.19] — The analysis estimated comparison of change from baseline to Week 48 between the DTG+RPV and CAR groups in total hip T-scores by baseline third agent NNRTI
Statistical Analysis 3: Comparison: DTG + RPV vs Current Antiretroviral Regimen; Test type: Other; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.09 to 0.24] — The analysis estimated comparison of change from baseline to Week 48 between the DTG+RPV and CAR groups in total hip T-scores by baseline third agent PI
Statistical Analysis 4: Comparison: DTG + RPV vs Current Antiretroviral Regimen; Test type: Other; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.25 to 0.37] — The analysis estimated comparison of change from baseline to Week 48 between the DTG+RPV and CAR groups in total hip Z-scores by baseline third agent INSTI
Statistical Analysis 5: Comparison: DTG + RPV vs Current Antiretroviral Regimen; Test type: Other; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [0.02 to 0.18] — The analysis estimated comparison of change from baseline to Week 48 between the DTG+RPV and CAR groups in total hip Z-scores by baseline third agent NNRTI
Statistical Analysis 6: Comparison: DTG + RPV vs Current Antiretroviral Regimen; Test type: Other; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.14 to 0.21] — The analysis estimated comparison of change from baseline to Week 48 between the DTG+RPV and CAR groups in total hip Z-scores by baseline third agent PI
Statistical Analysis 7: Comparison: DTG + RPV vs Current Antiretroviral Regimen; Test type: Other; Mean Difference (Final Values) = 0.36, 95% CI 2-sided [0.01 to 0.71] — The analysis estimated comparison of change from baseline to Week 48 between the DTG+RPV and CAR groups in lumbar spine T-scores by baseline third agent INSTI
Statistical Analysis 8: Comparison: DTG + RPV vs Current Antiretroviral Regimen; Test type: Other; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.03 to 0.25] — The analysis estimated comparison of change from baseline to Week 48 between the DTG+RPV and CAR groups in lumbar spine T-scores by baseline third agent NNRTI
Statistical Analysis 9: Comparison: DTG + RPV vs Current Antiretroviral Regimen; Test type: Other; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.30 to 0.33] — The analysis estimated comparison of change from baseline to Week 48 between the DTG+RPV and CAR groups in lumbar spine T-scores by baseline third agent PI
Statistical Analysis 10: Comparison: DTG + RPV vs Current Antiretroviral Regimen; Test type: Other; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [0.03 to 0.74] — The analysis estimated comparison of change from baseline to Week 48 between the DTG+RPV and CAR groups in lumbar spine Z-scores by baseline third agent INSTI
Statistical Analysis 11: Comparison: DTG + RPV vs Current Antiretroviral Regimen; Test type: Other; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.02 to 0.26] — The analysis estimated comparison of change from baseline to Week 48 between the DTG+RPV and CAR groups in lumbar spine Z-scores by baseline third agent NNRTI
Statistical Analysis 12: Comparison: DTG + RPV vs Current Antiretroviral Regimen; Test type: Other; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.26 to 0.34] — The analysis estimated comparison of change from baseline to Week 48 between the DTG+RPV and CAR groups in lumbar spine Z-scores by baseline third agent PI

10. Secondary Outcome: Percent Change From Baseline (Day 1) in Total Hip and Lumbar BMD by Baseline Third Agent-DTG+RPV Early Switch Group Through Early and Late Switch Phase
Description: Total hip and lumbar spine BMD (expressed as areal density in g/cm^2) assessed by third agent class (INSTI, NNRTI, PI) at indicated time points. Percent change from Baseline was calculated as post-dose value minus Baseline value divided by Baseline value multiplied by 100. BMD parameters expressed as areal density (g/cm^2) at Weeks 48, 100 and 148 reflect data adjusted following the ongoing longitudinal and cross-calibration of the multiple DEXA scanner instruments in this study. Data and analyses presented through Week 48 only represent the final results of Week 48 Primary Endpoint analysis which applied DEXA scanner calibrations though Week 48, with no subsequent calibration applied. In the final analysis conducted at Week 148, DEXA scanner calibration data acquired from Day 1 to Week 148 was applied to all raw DEXA BMD data at Weeks 48, 100 and 148. Hence, the actual values of Week 48 DEXA data may vary slightly between the Week 48 and Week 148 analyses.
Time Frame: Baseline (Day 1), Week 48, Week 100 and Week 148
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | DTG + RPV
Number analyzed (Participants) | 53
Percent change
  Total hip; INSTI; Week 48; n=7: number analyzed (Participants) | 7
  Total hip; INSTI; Week 48; n=7 | 1.918 (3.3468)
  Total hip; INSTI; Week 100; n=6: number analyzed (Participants) | 6
  Total hip; INSTI; Week 100; n=6 | 1.165 (4.5857)
  Total hip; INSTI; Week 148; n=6: number analyzed (Participants) | 6
  Total hip; INSTI; Week 148; n=6 | 1.738 (3.1881)
  Total hip; NNRTI; Week 48; n=28: number analyzed (Participants) | 28
  Total hip; NNRTI; Week 48; n=28 | 1.422 (2.4137)
  Total hip; NNRTI; Week 100; n=25: number analyzed (Participants) | 25
  Total hip; NNRTI; Week 100; n=25 | 0.722 (2.6977)
  Total hip; NNRTI; Week 148; n=24: number analyzed (Participants) | 24
  Total hip; NNRTI; Week 148; n=24 | 0.524 (4.0553)
  Total hip; PI; Week 48; n=11: number analyzed (Participants) | 11
  Total hip; PI; Week 48; n=11 | 1.401 (2.4406)
  Total hip; PI; Week 100; n=10: number analyzed (Participants) | 10
  Total hip; PI; Week 100; n=10 | 1.927 (3.7412)
  Total hip; PI; Week 148; n=10: number analyzed (Participants) | 10
  Total hip; PI; Week 148; n=10 | 1.610 (3.5534)
  Lumbar spine; INSTI; Week 48; n=7: number analyzed (Participants) | 7
  Lumbar spine; INSTI; Week 48; n=7 | 1.439 (2.2786)
  Lumbar spine; INSTI; Week 100; n=6: number analyzed (Participants) | 6
  Lumbar spine; INSTI; Week 100; n=6 | 0.779 (2.6627)
  Lumbar spine; INSTI; Week 148; n=6: number analyzed (Participants) | 6
  Lumbar spine; INSTI; Week 148; n=6 | -0.306 (0.8815)
  Lumbar spine; NNRTI; Week 48; n=28: number analyzed (Participants) | 28
  Lumbar spine; NNRTI; Week 48; n=28 | 1.570 (2.9752)
  Lumbar spine; NNRTI; Week 100; n=26: number analyzed (Participants) | 26
  Lumbar spine; NNRTI; Week 100; n=26 | -0.025 (3.9606)
  Lumbar spine; NNRTI; Week 148; n=25: number analyzed (Participants) | 25
  Lumbar spine; NNRTI; Week 148; n=25 | 0.067 (5.4222)
  Lumbar spine; PI; Week 48; n=11: number analyzed (Participants) | 11
  Lumbar spine; PI; Week 48; n=11 | 1.977 (2.5587)
  Lumbar spine; PI; Week 100; n=11: number analyzed (Participants) | 11
  Lumbar spine; PI; Week 100; n=11 | 2.801 (3.8743)
  Lumbar spine; PI; Week 148; n=11: number analyzed (Participants) | 11
  Lumbar spine; PI; Week 148; n=11 | 2.026 (3.8869)

11. Secondary Outcome: Change From Baseline (Day 1) in Total Hip and Lumbar Spine BMD T-scores and Z-scores by Baseline Third Agent-DTG+RPV Early Switch Group Through Early and Late Switch Phase
Description: T-score is the number of standard deviations above or below the mean BMD of a 30-year-old participant of same sex. Caucasian reference values were used to calculate T- and Z-scores. T-score values > -1.0 is normal; <= -1.0 to > -2.5 indicate osteopenia; <= -2.5 to <-3.5 indicate osteoporosis; <= -3.5 indicate severe osteoporosis. Z-score is the number of standard deviations above or below the mean BMD for a reference population of same age and sex in this study. Change from Baseline is the post-dose value minus Baseline value. Data for Week 48 only represents final results of Week 48 Primary Endpoint analysis which applied DEXA scanner calibrations through 48, with no subsequent calibration applied. In the final analysis conducted at Week 148, DEXA scanner calibration data acquired from Day 1 to Week 148 was applied to all raw DEXA BMD data at Weeks 48, 100 and 148. Hence, actual values of Week 48 DEXA data may vary slightly between Weeks 48 and 148 analyses.
Time Frame: Baseline (Day 1), Week 48, Week 100 and Week 148
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | DTG + RPV
Number analyzed (Participants) | 53
Scores on a scale
  INSTI; Total hip; T-score; Week 48; n=7: number analyzed (Participants) | 7
  INSTI; Total hip; T-score; Week 48; n=7 | 0.119 (0.2171)
  INSTI; Total hip; T-score; Week 100; n=6: number analyzed (Participants) | 6
  INSTI; Total hip; T-score; Week 100; n=6 | 0.069 (0.2854)
  INSTI; Total hip; T-score; Week 148; n=6: number analyzed (Participants) | 6
  INSTI; Total hip; T-score; Week 148; n=6 | 0.116 (0.2057)
  INSTI; Total hip; Z-score; Week 48; n=7: number analyzed (Participants) | 7
  INSTI; Total hip; Z-score; Week 48; n=7 | 0.162 (0.2402)
  INSTI; Total hip; Z-score; Week 100; n=6: number analyzed (Participants) | 6
  INSTI; Total hip; Z-score; Week 100; n=6 | 0.161 (0.2912)
  INSTI; Total hip; Z-score; Week 148; n=6: number analyzed (Participants) | 6
  INSTI; Total hip; Z-score; Week 148; n=6 | 0.219 (0.2360)
  INSTI; Lumbar spine; T-score; Week 48; n=7: number analyzed (Participants) | 7
  INSTI; Lumbar spine; T-score; Week 48; n=7 | 0.141 (0.2212)
  INSTI; Lumbar spine; T-score; Week 100; n=6: number analyzed (Participants) | 6
  INSTI; Lumbar spine; T-score; Week 100; n=6 | 0.087 (0.2611)
  INSTI; Lumbar spine; T-score; Week 148; n=6: number analyzed (Participants) | 6
  INSTI; Lumbar spine; T-score; Week 148; n=6 | -0.026 (0.0826)
  INSTI; Lumbar spine; Z-score; Week 48; n=7: number analyzed (Participants) | 7
  INSTI; Lumbar spine; Z-score; Week 48; n=7 | 0.196 (0.2100)
  INSTI; Lumbar spine; Z-score; Week 100; n=6: number analyzed (Participants) | 6
  INSTI; Lumbar spine; Z-score; Week 100; n=6 | 0.267 (0.3905)
  INSTI; Lumbar spine; Z-score; Week 148; n=6: number analyzed (Participants) | 6
  INSTI; Lumbar spine; Z-score; Week 148; n=6 | 0.191 (0.2644)
  NNRTI; Total hip; T-score; Week 48; n=28: number analyzed (Participants) | 28
  NNRTI; Total hip; T-score; Week 48; n=28 | 0.098 (0.1593)
  NNRTI; Total hip; T-score; Week 100; n=25: number analyzed (Participants) | 25
  NNRTI; Total hip; T-score; Week 100; n=25 | 0.045 (0.1938)
  NNRTI; Total hip; T-score; Week 148; n=24: number analyzed (Participants) | 24
  NNRTI; Total hip; T-score; Week 148; n=24 | 0.028 (0.2786)
  NNRTI; Total hip; Z-score; Week 48; n=28: number analyzed (Participants) | 28
  NNRTI; Total hip; Z-score; Week 48; n=28 | 0.107 (0.1574)
  NNRTI; Total hip; Z-score; Week 100; n=25: number analyzed (Participants) | 25
  NNRTI; Total hip; Z-score; Week 100; n=25 | 0.077 (0.1856)
  NNRTI; Total hip; Z-score; Week 148; n=24: number analyzed (Participants) | 24
  NNRTI; Total hip; Z-score; Week 148; n=24 | 0.071 (0.2958)
  NNRTI; Lumbar spine; T-score; Week 48; n=28: number analyzed (Participants) | 28
  NNRTI; Lumbar spine; T-score; Week 48; n=28 | 0.126 (0.2687)
  NNRTI; Lumbar spine; T-score; Week 100; n=26: number analyzed (Participants) | 26
  NNRTI; Lumbar spine; T-score; Week 100; n=26 | -0.022 (0.3558)
  NNRTI; Lumbar spine; T-score; Week 148; n=25: number analyzed (Participants) | 25
  NNRTI; Lumbar spine; T-score; Week 148; n=25 | -0.015 (0.4802)
  NNRTI; Lumbar spine; Z-score; Week 48; n=28: number analyzed (Participants) | 28
  NNRTI; Lumbar spine; Z-score; Week 48; n=28 | 0.150 (0.2669)
  NNRTI; Lumbar spine; Z-score; Week 100; n=26: number analyzed (Participants) | 26
  NNRTI; Lumbar spine; Z-score; Week 100; n=26 | 0.021 (0.3539)
  NNRTI; Lumbar spine; Z-score; Week 148; n=25: number analyzed (Participants) | 25
  NNRTI; Lumbar spine; Z-score; Week 148; n=25 | 0.049 (0.5248)
  PI; Total hip; T-Score; Week 48; n=11: number analyzed (Participants) | 11
  PI; Total hip; T-Score; Week 48; n=11 | 0.097 (0.1731)
  PI; Total hip; T-Score; Week 100; n=10: number analyzed (Participants) | 10
  PI; Total hip; T-Score; Week 100; n=10 | 0.118 (0.2740)
  PI; Total hip; T-Score; Week 148; n=10: number analyzed (Participants) | 10
  PI; Total hip; T-Score; Week 148; n=10 | 0.110 (0.2521)
  PI; Total hip; Z-Score; Week 48; n=11: number analyzed (Participants) | 11
  PI; Total hip; Z-Score; Week 48; n=11 | 0.106 (0.1823)
  PI; Total hip; Z-Score; Week 100; n=10: number analyzed (Participants) | 10
  PI; Total hip; Z-Score; Week 100; n=10 | 0.150 (0.2722)
  PI; Total hip; Z-Score; Week 148 ;n=10: number analyzed (Participants) | 10
  PI; Total hip; Z-Score; Week 148 ;n=10 | 0.166 (0.2441)
  PI; Lumbar spine; T-Score; Week 48 ;n=11: number analyzed (Participants) | 11
  PI; Lumbar spine; T-Score; Week 48 ;n=11 | 0.172 (0.2406)
  PI; Lumbar spine; T-Score; Week 100 ;n=11: number analyzed (Participants) | 11
  PI; Lumbar spine; T-Score; Week 100 ;n=11 | 0.235 (0.3396)
  PI; Lumbar spine; T-Score; Week 148 ;n=11: number analyzed (Participants) | 11
  PI; Lumbar spine; T-Score; Week 148 ;n=11 | 0.179 (0.3599)
  PI; Lumbar spine; Z-Score; Week 48 ;n=11: number analyzed (Participants) | 11
  PI; Lumbar spine; Z-Score; Week 48 ;n=11 | 0.257 (0.2601)
  PI; Lumbar spine; Z-Score; Week 100 ;n=11: number analyzed (Participants) | 11
  PI; Lumbar spine; Z-Score; Week 100 ;n=11 | 0.360 (0.3732)
  PI; Lumbar spine; Z-Score; Week 148 ;n=11: number analyzed (Participants) | 11
  PI; Lumbar spine; Z-Score; Week 148 ;n=11 | 0.317 (0.2828)

12. Secondary Outcome: Percent Change From LS Baseline (Week 48) Through Week 148 in Total Hip and Lumbar Spine BMD by Baseline Third Agent-CAR Late Switch Group Through Late Switch Phase
Description: Total hip and lumbar spine BMD (expressed as areal density in g/cm^2) assessed by third agent class (INSTI, NNRTI, PI) at indicated time points. The last pre-switch value (Week 48) was considered as LS Baseline and percent change from LS Baseline was calculated as post-dose value minus LS Baseline value divided by LS Baseline value multiplied by 100.
Time Frame: LS Baseline (Week 48), Week 100 and Week 148
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Current Antiretroviral Regimen
Number analyzed (Participants) | 44
Percent change
  Total hip; INSTI; Week 100; n=3: number analyzed (Participants) | 3
  Total hip; INSTI; Week 100; n=3 | 2.298 (2.7510)
  Total hip; INSTI; Week 148; n=3: number analyzed (Participants) | 3
  Total hip; INSTI; Week 148; n=3 | 2.405 (1.8787)
  Total hip; NNRTI; Week 100; n=29: number analyzed (Participants) | 29
  Total hip; NNRTI; Week 100; n=29 | 1.049 (2.9845)
  Total hip; NNRTI; Week 148; n=29: number analyzed (Participants) | 29
  Total hip; NNRTI; Week 148; n=29 | 1.498 (2.8487)
  Total hip; PI; Week 100; n=9: number analyzed (Participants) | 9
  Total hip; PI; Week 100; n=9 | 0.898 (1.7838)
  Total hip; PI; Week 148; n=8: number analyzed (Participants) | 8
  Total hip; PI; Week 148; n=8 | 0.042 (2.5640)
  Lumbar Spine; INSTI; Week 100; n=3: number analyzed (Participants) | 3
  Lumbar Spine; INSTI; Week 100; n=3 | 2.195 (1.1188)
  Lumbar Spine; INSTI; Week 148; n=3: number analyzed (Participants) | 3
  Lumbar Spine; INSTI; Week 148; n=3 | 1.121 (1.3711)
  Lumbar Spine; NNRTI; Week 100; n=29: number analyzed (Participants) | 29
  Lumbar Spine; NNRTI; Week 100; n=29 | 1.017 (2.7142)
  Lumbar Spine; NNRTI; Week 148; n=29: number analyzed (Participants) | 29
  Lumbar Spine; NNRTI; Week 148; n=29 | 0.335 (3.5996)
  Lumbar Spine; PI; Week 100; n=9: number analyzed (Participants) | 9
  Lumbar Spine; PI; Week 100; n=9 | 1.160 (5.1050)
  Lumbar Spine; PI; Week 148; n=8: number analyzed (Participants) | 8
  Lumbar Spine; PI; Week 148; n=8 | 0.546 (3.1654)

13. Secondary Outcome: Change From LS Baseline (Week 48) Through Week 148 in Total Hip and Lumbar Spine BMD T-scores and Z-scores by Baseline Third Agent-CAR Late Switch Group Through Late Switch Phase
Description: Total hip and lumbar spine BMD was assessed by Baseline third agent (INSTI, NNRTI, PI) using T-scores and Z-scores at indicated time points. DEXA scans of hip and spine were performed. The last pre-switch value (Week 48) was considered as LS Baseline and change from LS Baseline was calculated as the post-dose value minus LS Baseline value. T-score is the number of standard deviations above or below the mean BMD of a 30-year-old participant of the same sex. Caucasian reference values were used for all participants to calculate T-scores. T-score values > -1.0 are considered normal, T-score values <= -1.0 to > -2.5 indicate osteopenia, T-score values <= -2.5 to <-3.5 indicate osteoporosis and T-score values <= -3.5 indicate severe osteoporosis. The Z-score is the number of standard deviations above or below the mean BMD for a reference population of same age and sex and in this study. Caucasian reference values were used in calculation of Z-scores.
Time Frame: LS Baseline (Week 48), Week 100 and Week 148
Population: LS ITT-ED Population.Only those participants with data available at specified time point were analyzed (represented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Current Antiretroviral Regimen
Number analyzed (Participants) | 44
Scores on a scale
  INSTI; Hip; T-score; Week 100; n=3: number analyzed (Participants) | 3
  INSTI; Hip; T-score; Week 100; n=3 | 0.166 (0.1971)
  INSTI; Hip; T-score; Week 148; n=3: number analyzed (Participants) | 3
  INSTI; Hip; T-score; Week 148; n=3 | 0.173 (0.1333)
  INSTI; Hip; Z-score; Week 100; n=3: number analyzed (Participants) | 3
  INSTI; Hip; Z-score; Week 100; n=3 | 0.167 (0.1623)
  INSTI; Hip; Z-score; Week 148; n=3: number analyzed (Participants) | 3
  INSTI; Hip; Z-score; Week 148; n=3 | 0.197 (0.0800)
  INSTI; Spine; T-score; Week 100; n=3: number analyzed (Participants) | 3
  INSTI; Spine; T-score; Week 100; n=3 | 0.201 (0.1102)
  INSTI; Spine; T-score; Week 148; n=3: number analyzed (Participants) | 3
  INSTI; Spine; T-score; Week 148; n=3 | 0.099 (0.1164)
  INSTI; Spine; Z-score; Week 100; n=3: number analyzed (Participants) | 3
  INSTI; Spine; Z-score; Week 100; n=3 | 0.247 (0.0376)
  INSTI; Spine; Z-score; Week 148; n=3: number analyzed (Participants) | 3
  INSTI; Spine; Z-score; Week 148; n=3 | 0.145 (0.1888)
  NNRTI; Hip; T-score; Week 100; n=29: number analyzed (Participants) | 29
  NNRTI; Hip; T-score; Week 100; n=29 | 0.075 (0.2149)
  NNRTI; Hip; T-score; Week 148; n=29: number analyzed (Participants) | 29
  NNRTI; Hip; T-score; Week 148; n=29 | 0.106 (0.2064)
  NNRTI; Hip; Z-score; Week 100; n=29: number analyzed (Participants) | 29
  NNRTI; Hip; Z-score; Week 100; n=29 | 0.101 (0.2261)
  NNRTI; Hip; Z-score; Week 148; n=29: number analyzed (Participants) | 29
  NNRTI; Hip; Z-score; Week 148; n=29 | 0.136 (0.2213)
  NNRTI; Spine; T-score; Week 100; n=29: number analyzed (Participants) | 29
  NNRTI; Spine; T-score; Week 100; n=29 | 0.103 (0.2630)
  NNRTI; Spine; T-score; Week 148; n=29: number analyzed (Participants) | 29
  NNRTI; Spine; T-score; Week 148; n=29 | 0.045 (0.3441)
  NNRTI; Spine; Z-score; Week 100; n=29: number analyzed (Participants) | 29
  NNRTI; Spine; Z-score; Week 100; n=29 | 0.164 (0.2711)
  NNRTI; Spine; Z-score; Week 148; n=29: number analyzed (Participants) | 29
  NNRTI; Spine; Z-score; Week 148; n=29 | 0.124 (0.3482)
  PI; Hip; T-Score; Week 100; n=9: number analyzed (Participants) | 9
  PI; Hip; T-Score; Week 100; n=9 | 0.069 (0.1309)
  PI; Hip; T-Score; Week 148; n=8: number analyzed (Participants) | 8
  PI; Hip; T-Score; Week 148; n=8 | 0.007 (0.1856)
  PI; Hip; Z-Score; Week 100; n=9: number analyzed (Participants) | 9
  PI; Hip; Z-Score; Week 100; n=9 | 0.107 (0.1558)
  PI; Hip; Z-Score; Week 148 ;n=8: number analyzed (Participants) | 8
  PI; Hip; Z-Score; Week 148 ;n=8 | 0.061 (0.2111)
  PI; Spine; T-Score; Week 100 ;n=9: number analyzed (Participants) | 9
  PI; Spine; T-Score; Week 100 ;n=9 | 0.105 (0.4198)
  PI; Spine; T-Score; Week 148 ;n=8: number analyzed (Participants) | 8
  PI; Spine; T-Score; Week 148 ;n=8 | 0.044 (0.3052)
  PI; Spine; Z-Score; Week 100 ;n=9: number analyzed (Participants) | 9
  PI; Spine; Z-Score; Week 100 ;n=9 | 0.191 (0.2776)
  PI; Spine; Z-Score; Week 148 ;n=8: number analyzed (Participants) | 8
  PI; Spine; Z-Score; Week 148 ;n=8 | 0.133 (0.3817)

ADVERSE EVENTS:
Time Frame: On-treatment SAEs and non-serious AEs were collected from the start of the study treatment up to 148 weeks.
Description: AEs were reported for the Safety DEXA Population defined as participants in the parent Safety Populations who participated in the DEXA study. Only AEs considered related to the DEXA study procedure were collected in this study. All other AEs will be public disclosed for the parent studies (201636 [NCT02429791] and 201637 [NCT02422797]). Through the 148 weeks of conduct, no AEs considered related to the DEXA study procedure were reported. No deaths were reported for 202094 study participants.
Groups:
- DTG + RPV (Early Switch): Participants received DTG together with RPV once daily in an open-label fashion up to Week 52 during early switch phase in the parent study. Study medication was administered in the parent study (201636 [NCT02429791] and 201637 [NCT02422797]) and not in study 202094.
- CAR (Early Switch): Participants continued to receive their CAR (two NRTIs + a third agent). A third agent included either: an INSTI, a NNRTI or a PI. CAR was administered according to the approved labeling in an open-label fashion up to Week 52 during early switch phase in the parent study. Study medication was administered in the parent study (201636 [NCT02429791] and 201637 [NCT02422797]) and not in study 202094.
- DTG + RPV (Early + Late Switch): Participants received DTG together with RPV once daily in an open-label fashion up to Week 52 during early switch phase in the parent study and continued to receive DTG + RPV up to Week 148 during the Late Switch Phase in the parent study. Study medication was administered in the parent study (201636 [NCT02429791] and 201637 [NCT02422797]) and not in study 202094.
- CAR (Late Switch): At Week 52, participants who received CAR during the early switch phase, with HIV-1 RNA <50 c/mL, switched to DTG + RPV once daily and were followed until Week 148 in the parent study. Study medication was administered in the parent study (201636 [NCT02429791] and 201637 [NCT02422797]) and not in study 202094.
Arm/Group | DTG + RPV (Early Switch) | CAR (Early Switch) | DTG + RPV (Early + Late Switch) | CAR (Late Switch)
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/49 | 0/53 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/49 | 0/53 | 0/44
Other Adverse Events (participants affected / at risk) | 0/53 | 0/49 | 0/53 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.